CLINICAL TRIAL: NCT03283813
Title: Effects of a Supplementation With Zinc and Myo-inositol in Paediatric Obesity
Brief Title: ZIMBA: Clinical Trial in Paediatric Obesity
Acronym: ZIMBA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Azienda Ospedaliero Universitaria Maggiore della Carita (Other)
Responsible Party: Principal Investigator, Simonetta Bellone, Assoc. Professor, Azienda Ospedaliero Universitaria Maggiore della Carita
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CE 99/17
Record Dates: First submitted 2017-09-13; First posted 2017-09-14 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Obesity, Childhood; Insulin Resistance; Zinc Deficiency; Inositol
Keywords: Paediatric Obesity; Insulin resistance; Zinc; Myo-inositol
MeSH Terms: conditions — Pediatric Obesity; Insulin Resistance | interventions — Zinc; Inositol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The study is a triple blind study in which the treatment or intervention is unknown to the research participant, the individuals who administer the treatment or intervention, and the researchers who assess the outcomes.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active group - Zinc and Myo-inositol (Active Comparator): This arm will receive a supplementation with Zinc and Myo-inositol once a day.
  Interventions: Dietary Supplement: Zinc; Drug: Myoinositol
- Placebo group (Placebo Comparator): This arm will receive a supplementation with a same product equal to the active product but without Zinc and Myo-inositol inside.
  Interventions: Drug: Placebos

INTERVENTIONS:
Dietary Supplement: Zinc — In this active Group there will be a supplementation with Zinc (5 mg), Myo-inositol (2000 mg) and GOS (Galacto-oligosaccharides) of Pisum sativum (1000 mg)
  Arms: Active group - Zinc and Myo-inositol
Drug: Placebos — In this placebo Group there will be a supplementation with a product placebo equal to the active product with GOS (Galacto-oligosaccharides) of Pisum sativum(1000 mg) but without Zinc and Myo-inositol.
  Arms: Placebo group
Drug: Myoinositol — In this active Group there will be a supplementation with Zinc (5 mg), Myo-inositol (2000 mg) and GOS (Galacto-oligosaccharides) of Pisum sativum (1000 mg)
  Arms: Active group - Zinc and Myo-inositol

SUMMARY:
Myoinositol (MI) and D-chiro inositol (DCI) are isomeric forms of inositol that were found to have insulin-like properties, acting as second messengers in the insulin intracellular pathway; both of these molecules are involved in the increasing insulin sensitivity of different tissues to improve metabolic and ovulatory functions. Myoinositol is the predominant form that can be found in nature and food.

Inositol has been mainly used as a supplement in treating several pathologies such as polycystic ovary syndrome (PCOS), metabolic syndrome, type 2 diabetes mellitus (T2DM) and gestational diabetes (GDM). In the case of GDM, a condition defined as a glucose impairment first detected in pregnancy, a preventive role of inositol for GDM onset was recognized. In addition, inositol has been studied as a therapeutic option for the treatment of GDM and T2DM. The main effect of inositol is decreasing the level of insulin resistance. Consequently, a potential role of inositol as a treatment option could be hypothesized for other conditions typically characterized by insulin resistance like metabolic syndrome and obesity.

Zinc also plays an important role in insulin action and carbohydrate metabolism. It may also have a protective role in the prevention of atherogenesis. Several human studies have demonstrated that Zinc supplementation reduces total cholesterol, LDL cholesterol and triglycerides, in addition to increasing the HDL cholesterol levels. Studies have shown that diabetes is accompanied by hypozincemia and high levels of Zinc in urine. In addition Zinc is also an integral part of key anti-oxidant enzymes and Zinc deficiency impairs their synthesis, resulting in increased oxidative stress.

A supplementation with Myo-Inositol and Zinc could represent a valid strategy in paediatric obesity in addiction to a standard approach. The purpose of our study is to evaluate the supplementation of Myo-inositol and Zinc in the treatment of paediatric obesity.

DETAILED DESCRIPTION:
Study design: A single-center pilot open-label randomized control trial. Population: The study will comprise a total of 60 subjects of both sexes, with pubertal stage ≥ 3 according to the Tanner stage, obese according to the IOTF criteria (International Obesity Task Force), diet naïve or with failure of weight loss (defined as -1 kg/m2 BMI in 1 year).

Intervention: Patients will be randomized in a open-label, into two groups homogeneous for number and sex of the subjects. One group (group "active") will receive the supplementation with Myoinositol and Zinc (active product) and the other group (group "Placebo") will receive a placebo for a total of 3 months of treatment.

Dietary restriction: The standard diet will be distributed with 55-60% of carbohydrates, 25-30% lipids and 15% proteins, and will be performed in accordance with the calories of an isocaloric balanced diet calculated throughout the Italian LARN Guidelines for age and gender (Italian Society of Human Nutrition, 2014), inspired to Mediterranean pyramid.

Physical activity: all subjects will receive general recommendations about performing physical activity.

Randomization: Participants will be randomly assigned in a 1:1 to active intervention Group (Active Group) or Placebo Group.

Timing: Patients will be evaluated firstly at time of enrollment (V0) and at the end of the end of the study (V1).

The following anthropometric measures, biochemical and ultrasound evaluations and questionnaires will be obtained:

1. Anthropometric measures:

   * height (V0, V1);
   * weight (V0, V1);
   * body mass index (BMI; Kg/m2) (V0, V1);
   * waist and hip circumferences (V0, V1); for the calculation of the following ratios: waist/hip, waist/height;
   * Tanner stage (V0, V1); (Tanner JM, 1961);
   * blood pressure and heart rate (V0, V1);
2. Biochemical evaluations (after a 12-h overnight fast): CBC (Complete Blood Count) with formula, serum insulin-like growth factor 1 (IGF1, ng/mL), 25-hydroxy (OH) vitamin D (ng/mL), uric acid (mg/dL), Serum Zinc (mg/dl), alkaline phosphatase (U/L), ACTH (adrenocorticotropic hormone) (pg/mL), cortisol (microg/dL), TSH (thyroid-stimulating hormone)(uuI/mL), fT4 (serum free T4) (ng/dL) (V0, V1); aspartate aminotransferase (AST, IU/L), alanine aminotransferase (ALT, IU/L); AST-to-ALT ratio will be calculated as the ratio of AST (IU/L) and ALT(IU/L) (V0, V1); serum creatinine concentration (mg/dL) will be measured with the enzymatic method; according to the NKF-K/DOQI Guidelines for CKD in children and adolescents (Dialysis Outcome Quality Initiative), the eGFR will be calculated using updated Schwartz's formula: eGFR (mL/min/1.73 m2) = [0.413 x patient's height (cm)] / serum creatinine (mg/dL)(V0, V1); glucose (mg/dL), insulin (μUI/mL); insulin-resistance (IR) will be calculated using the formula of Homeostasis Model Assessment (HOMA)-IR: (insulin [mU/L] x glucose [mmol/lL) / 22.5)(V0, V1); lipid profile: total cholesterol (mg/dL), High-Density Lipoprotein (HDL)-cholesterol (mg/dL), triglycerides (mg/dL); Low-Density Lipoprotein (LDL)-cholesterol will be calculated by the Friedwald formula and non-HDL (nHDL)-cholesterol will be also calculated(V0, V1); oral glucose tolerance test (OGTT: 1.75 g of glucose solution per kg, maximum 75 g) and samples will be collected for the determination of glucose and insulin every 30 min. The area under the curve (AUC) for parameters after OGTT will be calculated according to the trapezoidal rule. Insulin sensitivity at fasting and during OGTT will be calculated as the formula of the Quantitative Insulin-Sensitivity Check Index (QUICKI) and Matsuda index (ISI). The insulinogenic index will be calculated as the ratio of the changes in insulin and glucose concentration from 0 to 30 min (InsI). Βeta-cell compensatory capacity will be evaluated by the disposition index defined as the product of the ISI and InsI (DI) (V0, V1); a collection at rest of first-morning urine sample. Physical and chemical urinalysis; urine albumin (mg/L) will be determined by an advanced immunoturbidimetric assay and urine creatinine (mg/dL) will be measured using the enzymatic method. Urine albumin to creatinine ratio (u-ACR - mg/g) (albumin-creatinine ratio), will be calculated using the following formula: [urine albumin (mg/dL) / urine creatinine (mg/dL)] x 1000. A sample of serum and a sample of plasma will be collected at each time and will be stocked in -20°C freezer for further laboratory analysis (V0, V1);
3. Nutritional and physical activity measurements:

   * KIDMED questionnaire for children and adolescents (Serra-Majem L et al., 2004). The Italian version is reported and approved by Istituto Superiore Sanità in Rapporti ISTISAN 12/42 (Istituto Superiore della Sanità, Rapporti ISTISAN 12/42, 2012)(V0, V1);
   * the Food Frequency Questionnaire section of the Children's Eating Habits Questionnaire (CEHQ-FFQ), performed by Identification and prevention of Dietary and lifestyle-induced health Effects In Children and infantS (IDEFICS) study (V0, V1);

Information retrieval: A case report form (CRF) will be completed for each subject included in the study. The source documents will be the hospital's or the physician's chart.

Statistical e sample size: A sample of 23 individuals has been estimated to be sufficient to demonstrate a difference of 2 points of HOMA-IR (Prodam F et al, 2013) with 90% power and a significance level of 95% and a drop-out rate of 10% using the Student test. Statistical significance will be assumed at P< 0.05. The statistical analysis will be performed with SPSS for Windows version 17.0 (SPSS Inc., Chicago, IL, USA).

Organization characteristics: The study will be conducted at the Pediatric Endocrine Service of Division of Pediatrics, Department of Health Sciences, University of Piemonte Orientale, in Novara.

All blood samples will be measured evaluated using standardized methods in the Hospital's Chemistry Laboratory, previously described (Prodam F et al., 2014 - Prodam F et al., 2016).

Good Clinical Practice: The protocol will be conducted in accordance with the declaration of Helsinki. Informed consent will be obtained from all parents.

ELIGIBILITY:
Inclusion Criteria:

* both sexes
* between 6 and 18 years of age
* obese, according to the IOTF criteria (Cole TJ et al., 2000)
* pubertal stage ≥ 3 according to the Tanner stage (Tanner et al., 1961)
* HOMA-IR > 2,5 or insulin > 15 µU/ml
* Serum Zinc level in the range of normality or under the normal levels.

Exclusion Criteria:

* Adverse reactions to the product or component of the product (allergies…)
* Genetic obesity (Prader Willi syndrome, Down syndrome), Metabolic obesity (Laurence-Biedl syndrome…), endocrinological obesity (Cushing syndrome, hypothyroidism)
* Chronic diseases, hepatic or gastroenterological diseases
* Medical treatment for chronic diseases
* Supplementation with inositol-like products or supplements containing Zinc and Inositol.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 56 (Actual)
Dates: Start 2018-02-05 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-03-10 (Actual)

PRIMARY OUTCOMES:
Change in HOMA-IR index | Change from baseline HOMA-IR (V0) at 3 months (V1).
  Evaluate if after the treatment with Myoinositol and Zinc supplementation there is a variation of HOMA-IR index.
  Evaluate if after the treatment with probiotic there is a variation of HOMA-IR index.

SECONDARY OUTCOMES:
Change in glucose level during oral glucose tolerance test (OGTT) | Change from Baseline OGTT (V0) at 3 months (V1)
  Evaluate if after the treatment with Myoinositol and Zinc supplementation there is a reduction of glucose values during the OGTT at time 0' e 120' after oral glucose tolerance test.
Metabolic control: Improvement of metabolic risk factors | Change from baseline lipid profile, insulin, leptin, adiponectin, GLP1 (V0) at 3 months (V1)
  Evaluate any variation of serum lipids, leptin, adiponectin, GLP1 and insulin during OGTT.

OTHER OUTCOMES:
Change in inflammatory cytokines. | Change from Baseline cytokines and metabolites (V0) at 3 months (V1).
  Evaluate new cytokines and metabolites that regulates hormone metabolism.

CONTACTS AND LOCATIONS:
Locations (1):
- AOU Maggiore della Carità - Clinica Pediatrica - Ambulatorio di Auxologia ed Endocrinologia Pediatrica, Novara, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Croze ML, Soulage CO. Potential role and therapeutic interests of myo-inositol in metabolic diseases. Biochimie. 2013 Oct;95(10):1811-27. doi: 10.1016/j.biochi.2013.05.011. Epub 2013 Jun 10. PMID 23764390
- [Background] Larner J. D-chiro-inositol--its functional role in insulin action and its deficit in insulin resistance. Int J Exp Diabetes Res. 2002;3(1):47-60. doi: 10.1080/15604280212528. PMID 11900279
- [Background] Genazzani AD, Lanzoni C, Ricchieri F, Jasonni VM. Myo-inositol administration positively affects hyperinsulinemia and hormonal parameters in overweight patients with polycystic ovary syndrome. Gynecol Endocrinol. 2008 Mar;24(3):139-44. doi: 10.1080/09513590801893232. PMID 18335328
- [Background] Muscogiuri G, Palomba S, Lagana AS, Orio F. Inositols in the Treatment of Insulin-Mediated Diseases. Int J Endocrinol. 2016;2016:3058393. doi: 10.1155/2016/3058393. Epub 2016 Sep 8. PMID 27688754
- [Background] Unfer V, Nestler JE, Kamenov ZA, Prapas N, Facchinetti F. Effects of Inositol(s) in Women with PCOS: A Systematic Review of Randomized Controlled Trials. Int J Endocrinol. 2016;2016:1849162. doi: 10.1155/2016/1849162. Epub 2016 Oct 23. PMID 27843451
- [Background] Corrado F, D'Anna R, Di Vieste G, Giordano D, Pintaudi B, Santamaria A, Di Benedetto A. The effect of myoinositol supplementation on insulin resistance in patients with gestational diabetes. Diabet Med. 2011 Aug;28(8):972-5. doi: 10.1111/j.1464-5491.2011.03284.x. PMID 21414183
- [Background] Pintaudi B, Di Vieste G, Bonomo M. The Effectiveness of Myo-Inositol and D-Chiro Inositol Treatment in Type 2 Diabetes. Int J Endocrinol. 2016;2016:9132052. doi: 10.1155/2016/9132052. Epub 2016 Oct 11. PMID 27807448
- [Background] Mancini M, Andreassi A, Salvioni M, Pelliccione F, Mantellassi G, Banderali G. Myoinositol and D-Chiro Inositol in Improving Insulin Resistance in Obese Male Children: Preliminary Data. Int J Endocrinol. 2016;2016:8720342. doi: 10.1155/2016/8720342. Epub 2016 Nov 1. PMID 27882052
- [Background] Marreiro DN, Fisberg M, Cozzolino SM. Zinc nutritional status and its relationships with hyperinsulinemia in obese children and adolescents. Biol Trace Elem Res. 2004 Aug;100(2):137-49. doi: 10.1385/bter:100:2:137. PMID 15326363
- [Background] Chausmer AB. Zinc, insulin and diabetes. J Am Coll Nutr. 1998 Apr;17(2):109-15. doi: 10.1080/07315724.1998.10718735. PMID 9550453
- [Background] Garg VK, Gupta R, Goyal RK. Hypozincemia in diabetes mellitus. J Assoc Physicians India. 1994 Sep;42(9):720-1. PMID 7883669
- [Background] Ranasinghe P, Pigera S, Galappatthy P, Katulanda P, Constantine GR. Zinc and diabetes mellitus: understanding molecular mechanisms and clinical implications. Daru. 2015 Sep 17;23(1):44. doi: 10.1186/s40199-015-0127-4. PMID 26381880
- [Background] Islam MR, Arslan I, Attia J, McEvoy M, McElduff P, Basher A, Rahman W, Peel R, Akhter A, Akter S, Vashum KP, Milton AH. Is serum zinc level associated with prediabetes and diabetes?: a cross-sectional study from Bangladesh. PLoS One. 2013 Apr 17;8(4):e61776. doi: 10.1371/journal.pone.0061776. Print 2013. PMID 23613929
- [Background] Jayawardena R, Ranasinghe P, Galappatthy P, Malkanthi R, Constantine G, Katulanda P. Effects of zinc supplementation on diabetes mellitus: a systematic review and meta-analysis. Diabetol Metab Syndr. 2012 Apr 19;4(1):13. doi: 10.1186/1758-5996-4-13. PMID 22515411
- [Background] Ranasinghe P, Wathurapatha WS, Ishara MH, Jayawardana R, Galappatthy P, Katulanda P, Constantine GR. Effects of Zinc supplementation on serum lipids: a systematic review and meta-analysis. Nutr Metab (Lond). 2015 Aug 4;12:26. doi: 10.1186/s12986-015-0023-4. eCollection 2015. PMID 26244049
- [Background] Kelishadi R, Hashemipour M, Adeli K, Tavakoli N, Movahedian-Attar A, Shapouri J, Poursafa P, Rouzbahani A. Effect of zinc supplementation on markers of insulin resistance, oxidative stress, and inflammation among prepubescent children with metabolic syndrome. Metab Syndr Relat Disord. 2010 Dec;8(6):505-10. doi: 10.1089/met.2010.0020. Epub 2010 Oct 28. PMID 21028969
- [Background] Serra-Majem L, Ribas L, Ngo J, Ortega RM, Garcia A, Perez-Rodrigo C, Aranceta J. Food, youth and the Mediterranean diet in Spain. Development of KIDMED, Mediterranean Diet Quality Index in children and adolescents. Public Health Nutr. 2004 Oct;7(7):931-5. doi: 10.1079/phn2004556. PMID 15482620
- [Background] Huybrechts I, Bornhorst C, Pala V, Moreno LA, Barba G, Lissner L, Fraterman A, Veidebaum T, Hebestreit A, Sieri S, Ottevaere C, Tornaritis M, Molnar D, Ahrens W, De Henauw S; IDEFICS Consortium. Evaluation of the Children's Eating Habits Questionnaire used in the IDEFICS study by relating urinary calcium and potassium to milk consumption frequencies among European children. Int J Obes (Lond). 2011 Apr;35 Suppl 1:S69-78. doi: 10.1038/ijo.2011.37. PMID 21483425
- [Background] Prodam F, Ricotti R, Genoni G, Parlamento S, Petri A, Balossini C, Savastio S, Bona G, Bellone S. Comparison of two classifications of metabolic syndrome in the pediatric population and the impact of cholesterol. J Endocrinol Invest. 2013 Jul-Aug;36(7):466-73. doi: 10.3275/8768. Epub 2012 Nov 27. PMID 23211535
- [Background] Tanner JM. (1961). Growth at adolescence. 2 edn. Oxford: Blackwell Scientific Publications.
- [Background] Cole TJ, Lobstein T. Extended international (IOTF) body mass index cut-offs for thinness, overweight and obesity. Pediatr Obes. 2012 Aug;7(4):284-94. doi: 10.1111/j.2047-6310.2012.00064.x. Epub 2012 Jun 19. PMID 22715120
- [Background] Società Italiana di Nutrizione Umana.(2014).Livelli di assunzione raccomandati di energia e nutrienti per la popolazione italiana (LARN). Milan, Italy: S.I.N.U.
- [Background] Cacciari E, Milani S, Balsamo A, Spada E, Bona G, Cavallo L, Cerutti F, Gargantini L, Greggio N, Tonini G, Cicognani A. Italian cross-sectional growth charts for height, weight and BMI (2 to 20 yr). J Endocrinol Invest. 2006 Jul-Aug;29(7):581-93. doi: 10.1007/BF03344156. PMID 16957405
- [Background] Kahn SE, Prigeon RL, McCulloch DK, Boyko EJ, Bergman RN, Schwartz MW, Neifing JL, Ward WK, Beard JC, Palmer JP, et al. Quantification of the relationship between insulin sensitivity and beta-cell function in human subjects. Evidence for a hyperbolic function. Diabetes. 1993 Nov;42(11):1663-72. doi: 10.2337/diab.42.11.1663. PMID 8405710
- [Background] Hogg RJ, Furth S, Lemley KV, Portman R, Schwartz GJ, Coresh J, Balk E, Lau J, Levin A, Kausz AT, Eknoyan G, Levey AS; National Kidney Foundation's Kidney Disease Outcomes Quality Initiative. National Kidney Foundation's Kidney Disease Outcomes Quality Initiative clinical practice guidelines for chronic kidney disease in children and adolescents: evaluation, classification, and stratification. Pediatrics. 2003 Jun;111(6 Pt 1):1416-21. doi: 10.1542/peds.111.6.1416. PMID 12777562
- [Background] Prodam F, Zanetta S, Ricotti R, Marolda A, Giglione E, Monzani A, Walker GE, Rampone S, Castagno M, Bellone S, Petri A, Aimaretti G, Bona G. Influence of Ultraviolet Radiation on the Association between 25-Hydroxy Vitamin D Levels and Cardiovascular Risk Factors in Obesity. J Pediatr. 2016 Apr;171:83-9.e1. doi: 10.1016/j.jpeds.2015.12.032. Epub 2016 Jan 12. PMID 26794470
- [Background] Prodam F, Savastio S, Genoni G, Babu D, Giordano M, Ricotti R, Aimaretti G, Bona G, Bellone S. Effects of growth hormone (GH) therapy withdrawal on glucose metabolism in not confirmed GH deficient adolescents at final height. PLoS One. 2014 Jan 30;9(1):e87157. doi: 10.1371/journal.pone.0087157. eCollection 2014. PMID 24498035
- [Background] Cook S, Weitzman M, Auinger P, Nguyen M, Dietz WH. Prevalence of a metabolic syndrome phenotype in adolescents: findings from the third National Health and Nutrition Examination Survey, 1988-1994. Arch Pediatr Adolesc Med. 2003 Aug;157(8):821-7. doi: 10.1001/archpedi.157.8.821. PMID 12912790
- [Background] de Ferranti SD, Gauvreau K, Ludwig DS, Neufeld EJ, Newburger JW, Rifai N. Prevalence of the metabolic syndrome in American adolescents: findings from the Third National Health and Nutrition Examination Survey. Circulation. 2004 Oct 19;110(16):2494-7. doi: 10.1161/01.CIR.0000145117.40114.C7. Epub 2004 Oct 11. PMID 15477412
- [Background] Cruz ML, Goran MI. The metabolic syndrome in children and adolescents. Curr Diab Rep. 2004 Feb;4(1):53-62. doi: 10.1007/s11892-004-0012-x. PMID 14764281